CLINICAL TRIAL: NCT01431872
Title: Systemic DKK1 During Estrogen Level Changes in Post-menopausal Breast Cancer Patients Treated With Aromatase Inhibitors
Brief Title: Systemic Dickkopf-related Protein 1 (DKK1)During Estrogen Level Changes in Post-menopausal Breast Cancer Patients Treated With Aromatase Inhibitors
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 131471
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post menopausal breast cancer patients

SUMMARY:
The investigators are hypothesizing that decreasing estrogen levels will cause serum DKK1 to peak, then decrease gradually as estrogens reach a new lower, but steady level. The investigators also believe that the peak in DKK1 will initiated a wave of stem cell diversion from the osteoblastogenic pathway to the adipogenic pathway.

The investigators will conduct a longitudinal cohort study of post menopausal women with hormone-responsive breast cancer that will be treated AIs. The study will observe anthromorphic and serum marker changes during the first year of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Post Menopausal Breast cancer patients with planned treatment of aromatase inhibitors.
* 18 years or older

Exclusion Criteria:

* BMI >30 or <18
* Osteoporosis as defined by protocol.
* Subjects currently on bisphosphonate therapy.
* History of primary or secondary hyperparathyroidism
* History of Hypo-or Hyperthyroidism
* History of Vitamin D levels below LLN
* History of creatinine clearance below the EGFR
* History ofLiver function tests above 1.5 times ULN including LDH, SGOT, SGPT, Alkaline phosphatase, and Bilirubin
* History of documented cirrhosis of the liver
* History of chronic heparin use
* History of chronic glucocorticoid therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post menopausal breast cancer patients who are planning to be treated with aromatase inhibitors.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Estrogen level suppresses DKK1 | 26 weeks
  With the start of AI treatment, estrogen levels will decline to almost undetectable levels. We believe this decrease in estrogen will lift suppression of DKK1 and allow its expression to peak during the 1st month of treatment, and decline more slowly thereafter. During the first 26 weeks of treatment, we expect levels of CTx to rise, PTH to fall, and P1NP to show no change, findings that would be consistent with Heshmati's study.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hutchins, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States